CLINICAL TRIAL: NCT03699605
Title: Development and Feasibility Analysis of Verbal Expressive Skills Management Programme (VESMP) for Patients With Broca Aphasia
Acronym: VESMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Humaira Shamim, Assistant Professor, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIRS-IUISB/PHD/015
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Aphasia, Broca; Stroke
Keywords: Stroke; Aphasia; Broca Aphasia; communication skills; Verbal expressive skill management programme
MeSH Terms: conditions — Aphasia, Broca; Stroke; Aphasia

STUDY DESIGN:
Intervention Model Description: The two groups were included for speech therapy. For any given subject, aphasia severity evaluations were completed on the same day.includes patients that are 40+ years old, and have three months of post stroke with diagnosis of chronic Broca's Aphasias, each patient received treatment for 4 months that includes 04 VESMP sessions per week with each session being 30-45 minutes long. The measurement will be taken at 0 week (baseline) after 16 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VESMP (Experimental): Participants used VESMP at least half hour session thrice a week over an average of 4 months. The instruction before every domain included using it independently on the participant's own smart phone, or with a trained person either in the clinic or on their phone brought to the participant's home.
  Total 25 patients with diagnosis of severe non-fluent aphasia included, ages 40+, at least 3 months post-onset of single unilateral CVA affecting the language dominant hemisphere at the time of baseline testing also including, Participant demographics, aphasia classification and severity. All subjects participated in an intensive 2-week VESMP treatment program prior to beginning the individualized programs.
  Interventions: Other: VESMP
- Traditional Therapy (Active Comparator): Control group received traditional therapy total 25 patients with diagnosis of severe non-fluent aphasia included, All subjects participated in an traditional therapy group in routine and received language therapy for 4 months of periods with three sessions per week.
  Interventions: Other: Traditional Therapy

INTERVENTIONS:
Other: VESMP — . The application contains following seven domains: spontaneous speech, comprehension, naming, reading, writing, imitation and automated speech. The programme was developed in Urdu language which contains different daily functional words, phrases and sentences. Treatment stimuli consisted of images of objects along with auditory sounds of person and actions cues. The voice output can operate by pressing the selected picture with index finger. Participants received 1-16 weeks of therapy using software of two domains with different difficulty levels. Specifically the programme included seven domains within the software comprising of eight 30-45 minutes sessions (4 days per week for total 16weeks). The measurement will be taken at 0 week (baseline) after 16 weeks.
  Arms: VESMP
Other: Traditional Therapy — , All subjects participated in an traditional therapy group in routine and received MIT for 4 months of periods with three sessions per week to improve language skills.
  Other Names: MIT
  Arms: Traditional Therapy

SUMMARY:
The present study was conducted to develop the verbal expressive skills management programme (VESMP) to enhance verbal expressive skills of patients with severe Broca aphasia. To determine the efficacy of VESMP in improving the quality of life and level of satisfaction of aphasic stroke patients.Control group received traditional therapy and experimental group received therapy through VESMP programme on their smart phones.

DETAILED DESCRIPTION:
Speech therapy makes an integral part of the non-pharmacological, conservative management of Post stroke aphasia. Routine speech therapy aims to improve comprehension and verbal skills and also develop functional communication skills through augmentative Alternative communication devices. Disorders of communication, including aphasia (mainly post stroke) caused by the left hemisphere brain damage, is a major community health issue. Aphasia is a language disorder occurring mainly as a result of stroke. It is an acquired impairment of language that weakens people's ability of comprehension and expression, it does not show any affect to intellect ability. The verbal expressive skills management programme (VESMP) is the software which developed augmented management for patients to enhance verbal expressive skills for patients with severe Broca's aphasia from different geographic areas.

ELIGIBILITY:
Inclusion Criteria:

* The 40-60 year Broca aphasia patients
* The severe Broca aphasia patients (more than 03 month of onset of stroke) Both infarct and hemorrhagic stroke
* Either gender Informed consent

Exclusion Criteria:

* • Broca Aphasic patients having cognitive impairment

  * The patients having tumors, infections and trauma

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Boston Diagnostic Aphasia Examination Battery (BDAE) | 16 weeks
  The Boston Diagnostic Aphasia Examination Battery (BDAE) was administered to all participants pre-and post-VESMP. The BDAE is a comprehensive standardized test of language performance for individuals with aphasia that includes measures of spoken language, naming, auditory comprehension, reading and other modalities.
Stroke Quality of life Scale | 16 weeks
  Scoring: each item shall be scored with the following key Total help - Couldn't do it at all - Strongly agree 1 A lot of help - A lot of trouble - Moderately agree 2 Some help - Some trouble - Neither agree nor disagree 3 A little help - A little trouble - Moderately disagree 4 No help needed - No trouble at all - Strongly disagree 5

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Railway Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Kiyani HS, Naz S, Mubeen R, Zubair R. Effectiveness of a Verbal Expressive Skills Management Program for Pakistani Patients with Broca Aphasia: A Randomized Clinical Trial. Altern Ther Health Med. 2023 Sep;29(6):204-208. PMID 37295011